CLINICAL TRIAL: NCT05557279
Title: Urinary Microbiome Changes Following Administration of 500 mg of NDS-446 in Women With Dry OAB at 12 Weeks - a Single-center Study
Brief Title: Urinary Microbiome Changes Following Administration of 500 mg of NDS-446 in Women With Dry OAB at 12 Weeks
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Elizabeth Mueller MD, Principal Investigator, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215838
Record Dates: First submitted 2022-09-12; First posted 2022-09-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: All participants will receive 500 mg NDS-446 daily for 12 weeks following a baseline assessment and meeting inclusion/exclusion criteria 20 premenopausal women, 20 postmenopausal women not on estrogen supplementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Other): All participants will receive 500 mg NDS-446 daily for 12 weeks
  Interventions: Drug: 500 mg NDS-446

INTERVENTIONS:
Drug: 500 mg NDS-446 — All participants will receive 500 mg NDS-446 daily for 12 weeks following a baseline assessment

SUMMARY:
The purpose of this study is to learn about how the use of 500 mg of dried cranberry powder extract (NDS-446) changes the bacteria that normal reside in the bladder of women who don't have urinary leakage problems but do have problems with urinary urgency and frequency.

DETAILED DESCRIPTION:
While this treatment algorithm is the recommended approach to OAB management, recent research has resulted in the development of a new paradigm that may influence how this condition is treated in the future. This research focuses on the urinary microbiome and for a decade it has been known that urine is not sterile. Expanded Quantitative Urine Culture (EQUC) techniques have allowed for more comprehensive and accurate 16S ribosomal RNA sequencing of the urinary microbiome. Changes in the abundance and diversity of the resident microbiota have been associated with a number of urogenital conditions including interstitial cystitis, urinary incontinence, responses to OAB medications and symptoms of urinary tract infections. These studies provide insight to the fact that the microbiome plays an important role in the maintenance of a healthy urogenital tract. Thus, treatments that target the microbiome for one condition may work for others by similar mechanisms, especially when there is considerable symptom overlap between the two conditions as there is in UTIs and OAB.

One such treatment is cranberry (Vaccinium macrocarpon) extract, which has long been used as complementary therapy for a variety of medical conditions. Health benefits are linked to the presence of phytochemicals present in the fruit- anthocyanins, flavonols, tannins, proanthocyanidins, and phenolic acid derivatives. Cranberry is known to be effective in the prevention of UTIs. In a recent study examining its use in women with dry OAB, daily dried cranberry improved urgency symptoms and number of daytime voids. In addition, the authors reported an improvement in the validated subjective instrument, Patient Perception of Bladder Condition (PPBC). Moderately symptomatic LUTS in men improved following 6 months of daily dried cranberry powder. Therefore, the investigators aim to investigate changes to the female urinary microbiome in women with dry OAB who take daily dried cranberry extract. This study aims to quantify a change in urinary frequency, urinary urgency, and PPBC following the daily use of a cranberry extract called NDS-446. The investigators also have an ancillary hypothesis that women who are post-menopausal will develop a urinary microbiome more similar to pre-menopausal women by the end of the study. Lastly, the investigators will measure the levels of extracellular (eATP) in the urine of participants. It has been previously shown that higher levels of eATP are associated with worsening OAB symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years, female, ambulatory
* OAB symptoms > 6 months
* Voiding frequency > 8 times in 24 hrs and > 3 episodes of urgency (grade 3 or 4) without incontinence during 3-day diary at baseline

Exclusion Criteria:

* Self-reported urinary incontinence (> 3 episodes in the month prior)
* UTI > 3 in last 12 months
* A diagnosis of painful bladder syndrome or interstitial cystitis
* LUT surgery last 6 months
* Drug or non-drug treatment of OAB (previous 60 days) or current meds that affect detrusor activity
* On Warfarin
* Failure to complete 3-day diary
* Aspirin > 81 mg daily
* Gross hematuria
* Allergy or sensitivity to aspirin
* Subjects taking anti-platelet agents
* Inability to swallow capsules

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Compare the UG microbiota (vagina, peri-urethral, catheterized and voided urine) of female participants with urgency-frequency syndrome after 12 weeks of daily use of 500 mg of NDS-446 to the UG microbiota at baseline. | 12 week visit
  Vaginal and peri-urethral swabs, as well as voided and catheterized urine specimens, will be obtained.

SECONDARY OUTCOMES:
Compare the baseline and 12 week PPBC score in pre-menopausal and post-menopausal who take 500 mg of NDS-446 daily. | 12 week visit
  The Patient Perception of Bladder Condition (PPBC) score in the study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mueller, MD, Principal Investigator — Loyola Medical Center
Locations (1):
- Loyola Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Milsom I, Kaplan SA, Coyne KS, Sexton CC, Kopp ZS. Effect of bothersome overactive bladder symptoms on health-related quality of life, anxiety, depression, and treatment seeking in the United States: results from EpiLUTS. Urology. 2012 Jul;80(1):90-6. doi: 10.1016/j.urology.2012.04.004. PMID 22748867
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] Madhuvrata P, Cody JD, Ellis G, Herbison GP, Hay-Smith EJ. Which anticholinergic drug for overactive bladder symptoms in adults. Cochrane Database Syst Rev. 2012 Jan 18;1:CD005429. doi: 10.1002/14651858.CD005429.pub2. PMID 22258963
- [Background] Coupland CAC, Hill T, Dening T, Morriss R, Moore M, Hippisley-Cox J. Anticholinergic Drug Exposure and the Risk of Dementia: A Nested Case-Control Study. JAMA Intern Med. 2019 Aug 1;179(8):1084-1093. doi: 10.1001/jamainternmed.2019.0677. PMID 31233095
- [Background] Chapple CR, Nazir J, Hakimi Z, Bowditch S, Fatoye F, Guelfucci F, Khemiri A, Siddiqui E, Wagg A. Persistence and Adherence with Mirabegron versus Antimuscarinic Agents in Patients with Overactive Bladder: A Retrospective Observational Study in UK Clinical Practice. Eur Urol. 2017 Sep;72(3):389-399. doi: 10.1016/j.eururo.2017.01.037. Epub 2017 Feb 11. PMID 28196724
- [Background] Wolfe AJ, Toh E, Shibata N, Rong R, Kenton K, Fitzgerald M, Mueller ER, Schreckenberger P, Dong Q, Nelson DE, Brubaker L. Evidence of uncultivated bacteria in the adult female bladder. J Clin Microbiol. 2012 Apr;50(4):1376-83. doi: 10.1128/JCM.05852-11. Epub 2012 Jan 25. PMID 22278835
- [Background] Siddiqui H, Nederbragt AJ, Lagesen K, Jeansson SL, Jakobsen KS. Assessing diversity of the female urine microbiota by high throughput sequencing of 16S rDNA amplicons. BMC Microbiol. 2011 Nov 2;11:244. doi: 10.1186/1471-2180-11-244. PMID 22047020
- [Background] Price TK, Dune T, Hilt EE, Thomas-White KJ, Kliethermes S, Brincat C, Brubaker L, Wolfe AJ, Mueller ER, Schreckenberger PC. The Clinical Urine Culture: Enhanced Techniques Improve Detection of Clinically Relevant Microorganisms. J Clin Microbiol. 2016 May;54(5):1216-22. doi: 10.1128/JCM.00044-16. Epub 2016 Mar 9. PMID 26962083
- [Background] Brubaker L, Nager CW, Richter HE, Visco A, Nygaard I, Barber MD, Schaffer J, Meikle S, Wallace D, Shibata N, Wolfe AJ. Urinary bacteria in adult women with urgency urinary incontinence. Int Urogynecol J. 2014 Sep;25(9):1179-84. doi: 10.1007/s00192-013-2325-2. Epub 2014 Feb 11. PMID 24515544
- [Background] Burnett LA, Hochstedler BR, Weldon K, Wolfe AJ, Brubaker L. Recurrent urinary tract infection: Association of clinical profiles with urobiome composition in women. Neurourol Urodyn. 2021 Aug;40(6):1479-1489. doi: 10.1002/nau.24707. Epub 2021 May 26. PMID 34036621
- [Background] Pearce MM, Zilliox MJ, Rosenfeld AB, Thomas-White KJ, Richter HE, Nager CW, Visco AG, Nygaard IE, Barber MD, Schaffer J, Moalli P, Sung VW, Smith AL, Rogers R, Nolen TL, Wallace D, Meikle SF, Gai X, Wolfe AJ, Brubaker L; Pelvic Floor Disorders Network. The female urinary microbiome in urgency urinary incontinence. Am J Obstet Gynecol. 2015 Sep;213(3):347.e1-11. doi: 10.1016/j.ajog.2015.07.009. Epub 2015 Jul 23. PMID 26210757
- [Background] Thomas-White KJ, Hilt EE, Fok C, Pearce MM, Mueller ER, Kliethermes S, Jacobs K, Zilliox MJ, Brincat C, Price TK, Kuffel G, Schreckenberger P, Gai X, Brubaker L, Wolfe AJ. Incontinence medication response relates to the female urinary microbiota. Int Urogynecol J. 2016 May;27(5):723-33. doi: 10.1007/s00192-015-2847-x. Epub 2015 Sep 30. PMID 26423260
- [Background] Jepson RG, Williams G, Craig JC. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD001321. doi: 10.1002/14651858.CD001321.pub5. PMID 23076891
- [Background] Cho A, Eidelberg A, Butler DJ, Danko D, Afshinnekoo E, Mason CE, Chughtai B. Efficacy of Daily Intake of Dried Cranberry 500 mg in Women with Overactive Bladder: A Randomized, Double-Blind, Placebo Controlled Study. J Urol. 2021 Feb;205(2):507-513. doi: 10.1097/JU.0000000000001384. Epub 2020 Sep 18. PMID 32945735
- [Background] Vidlar A, Student V Jr, Vostalova J, Fromentin E, Roller M, Simanek V, Student V. Cranberry fruit powder (Flowens) improves lower urinary tract symptoms in men: a double-blind, randomized, placebo-controlled study. World J Urol. 2016 Mar;34(3):419-24. doi: 10.1007/s00345-015-1611-7. Epub 2015 Jun 7. PMID 26049866
- [Background] Vidlar A, Vostalova J, Ulrichova J, Student V, Stejskal D, Reichenbach R, Vrbkova J, Ruzicka F, Simanek V. The effectiveness of dried cranberries ( Vaccinium macrocarpon) in men with lower urinary tract symptoms. Br J Nutr. 2010 Oct;104(8):1181-9. doi: 10.1017/S0007114510002059. Epub 2010 Aug 31. PMID 20804630
- [Background] Silva-Ramos M, Silva I, Oliveira O, Ferreira S, Reis MJ, Oliveira JC, Correia-de-Sa P. Urinary ATP may be a dynamic biomarker of detrusor overactivity in women with overactive bladder syndrome. PLoS One. 2013 May 31;8(5):e64696. doi: 10.1371/journal.pone.0064696. Print 2013. PMID 23741373
- [Background] Thomas-White K, Taege S, Limeira R, Brincat C, Joyce C, Hilt EE, Mac-Daniel L, Radek KA, Brubaker L, Mueller ER, Wolfe AJ. Vaginal estrogen therapy is associated with increased Lactobacillus in the urine of postmenopausal women with overactive bladder symptoms. Am J Obstet Gynecol. 2020 Nov;223(5):727.e1-727.e11. doi: 10.1016/j.ajog.2020.08.006. Epub 2020 Aug 11. PMID 32791124
- [Background] Price TK, Wolff B, Halverson T, Limeira R, Brubaker L, Dong Q, Mueller ER, Wolfe AJ. Temporal Dynamics of the Adult Female Lower Urinary Tract Microbiota. mBio. 2020 Apr 21;11(2):e00475-20. doi: 10.1128/mBio.00475-20. PMID 32317321
- [Background] Coyne KS, Matza LS, Kopp Z, Abrams P. The validation of the patient perception of bladder condition (PPBC): a single-item global measure for patients with overactive bladder. Eur Urol. 2006 Jun;49(6):1079-86. doi: 10.1016/j.eururo.2006.01.007. Epub 2006 Jan 24. PMID 16460875
- [Background] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047
- [Background] Gao X, Lin H, Revanna K, Dong Q. A Bayesian taxonomic classification method for 16S rRNA gene sequences with improved species-level accuracy. BMC Bioinformatics. 2017 May 10;18(1):247. doi: 10.1186/s12859-017-1670-4. PMID 28486927
- [Background] McMurdie PJ, Holmes S. Phyloseq: a bioconductor package for handling and analysis of high-throughput phylogenetic sequence data. Pac Symp Biocomput. 2012:235-46. PMID 22174279